CLINICAL TRIAL: NCT01235143
Title: Comparison the Incidence of Emergence Agitation Between Sevoflurane and Desflurane After Pediatric Urologic Surgery
Brief Title: Emergence Agitation Between Sevoflurane and Desflurane in Pediatric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, maliwan oofuvong, Assistant Professor, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PSU 136
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Children; Urologic Diseases; Ambulation Difficulty
Keywords: incidence; emergence agitation; sevoflurane; desflurane; ambulatory pediatric surgery
MeSH Terms: conditions — Urologic Diseases; Mobility Limitation; Emergence Delirium | interventions — Desflurane; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- desflurane anesthesia (Experimental): maintenance anesthesia with desflurane
  Interventions: Drug: Desflurane
- sevoflurane (Active Comparator): maintenance anesthesia with sevoflurane
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Desflurane — Desflurane (not more than 1 MAC) for maintenance of anesthesia in urologic surgery
  Other Names: Suprane (desflurane, USP)
  Arms: desflurane anesthesia
Drug: Sevoflurane — Sevoflurane (not more than 1 MAC) for maintenance of anesthesia in urologic surgery
  Other Names: sevorane
  Arms: sevoflurane

SUMMARY:
Sevoflurane is the volatile anesthetic agent of choice in pediatric surgery. Nevertheless, sevoflurane anesthesia had the high incidence of emergence delirium compared to halothane and isoflurane.Bortone L et al.reported isoflurane for maintenance decreased incidence of emergence agitation compared to sevoflurane in unpremedicated preschool children under elective subumbilical surgery (32% versus 52% respectively). Desflurane is the new volatile anesthetic agent which provides faster recovery compared to sevoflurane.Valley et al.reported no significant differences between sevoflurane or desflurane anesthesia in children in term of the serious airway complication such as laryngospasm or desaturation excepted the number of coughing episodes were more frequent in the desflurane compared to sevoflurane (36 versus 18).Mayer J et al. reported sevoflurane had severity of Pediatric Anesthesia Emergence Delirium (PAED) scale higher than desflurane in ear, nose, throat inpatient surgery in children (12(2-20) versus 6(0-15) respectively) with no reported of incidence of emergence agitation between those two. Therefore, the investigators would like to compare the incidence of emergence agitation, recovery profile and respiratory events between desflurane and sevoflurane anesthesia in pediatric ambulatory urologic surgery under general anesthesia and combined with regional anesthesia.

DETAILED DESCRIPTION:
After institutional review board (Prince of Songkla University, Songkhla, Thailand) approval and written informed consent from parents, 136 children aged 1-9 years, with American Society of Anesthesiologists (ASA) physical status I or II ,scheduled to undergoing elective ambulatory urologic surgery under general anesthesia combined with regional block , were prospectively enrolled in the study. Children were randomized by a computer-generated program to either sevoflurane group (group s, n =68) or desflurane group (group d, n =68) for maintenance of anesthesia . Exclusion criterion included emergency procedures, medical contraindication to placement of a caudal block, mental retardation, developmental delay, attention-deficit/hyperactivity disorder, psychiatric illness, a history of paradoxical excitation with sedatives. Children did not receive any premedication. Parents were allowed to be present for induction. Children's behavior was assessed at the time of separation from parents by using a separation scale 1-4 (1= excellent [separates easily] , 2= good [not clinging, whimpers ,calm with reassurance] , 3 = fair [not clinging , cried , will not calm or quiet] , 4 = poor [crying , clinging to parent]11 . A separation score of 1 or 2 was considered satisfactory , whereas a score of 3 or 4 was considered unsatisfactory. An induction scale 1-4 was used to assess acceptance of the anesthetic mask ( 1 = excellent [unafraid, co-operate, accepts mask readily], 2 = good [slight fear of mask , easily calmed] , 3 = fair[ moderated fear , not calmed with reassurance] ,4 = poor [terrified , crying ,agitated]11. An induction score of 1 or 2 was considered satisfactory , whereas a score of 3 or 4 was considered unsatisfactory. Then , children received a mask induction with either incremental sevoflurane 2-8% or single breath sevoflurane 8% in a 70 % nitrous oxide and 30% oxygen mixture with a 10 L/min fresh gas flow. After inhalation anesthetic induction , an intravenous cannula were place. Ventilation was controlled by laryngeal mask airway (LMA). After established the airway, children were assigned to receive either sevoflurane or desflurane by adjusting end-tidal concentration to deliver a minimum alveolar anesthetic concentration(MAC) of 1. The nitrous oxide in oxygen concentration was reduced to 66% and total gas flow rate was reduced to 5 LMP . All regional block; penile block, ilioinguinal nerve block and caudal block , were performed by discretion of attending anesthesiologist based on routine practice and type of operation.

Intraoperative analgesics or other sedative drug were not given unless the child's heart rate increase > 20% of baseline after incision or during operation and then fentanyl 0.5-1 mcg/kg intravenously was given to supplement analgesia throughout the operation. At the start of surgical closure, the inhaled anesthetic was discontinued. When the wound closure was completed , the nitrous oxide was discontinued with the oxygen flow rate was increase to 10 LMP. The awake LMA removal was followed by extubation criteria. The children were then transported to the post-anesthetic care unit (PACU). The awakening time defined by the time after discontinued inhaled agent until LMA was removed. Duration of surgery and anesthesia were also recorded. The emergence agitation score was assessed by 3 experienced PACU nurse, blinded to the inhaled anesthetic agents. The emergence agitation score 1-4 and duration of agitation were measured in the PACU (1= awake and calm , cooperative ; 2 = crying, requires consoling ; 3 = irritable/restless , screaming , inconsolable ; 4 = combative ,disoriented, thrashing)11. Children with an agitation score of 3 or 4 were classified agitated. Parent were reunited with their children in the PACU after an initial admission and stabilization phase. The pain score 1-10 using the FLACC under the age of 5 and the Face Pain Scale or the Numeric Rating Scale in older children was assessed by the same PACU nurse. If the children had severely agitated by agitation score > 3 for 5 minutes or pain score ≥ 4, the fentanyl 0.5 mcg/kg was administered intravenously every 10-15 min for treatment of agitation or rescue analgesia. Maximum agitation score and maximum pain score were recorded in the PACU. Duration in PACU stay defined by the time arrived in the PACU until discharge from PACU were also recorded. Intraoperative respiratory adverse events and PACU adverse events were recorded.

Primary objective was to compare the incidence of emergence agitation between sevoflurane anesthesia and desflurane anesthesia in pediatric ambulatory urologic surgery. Secondary objectives were to compare the recovery profile such as awakening time. Duration of PACU stay, and also intraoperative and PACU respiratory adverse events between sevoflurane anesthesia and desflurane anesthesia.

The statistic analysis The sample size calculation by program R 2.8.1 was based on the incidence of sevoflurane induced emergence agitation 52% by Bortone, et al 4 . the investigators calculated a sample size of 62 subjects per treatment arm wound have at least an 80% power to detect desflurane reduced of 50% compared to sevoflurane in the incidence of emergency agitation. The calculation was included the 10% dropout of the study, so 136 children were enrolled in the study.

Date were reported as mean±SD , median (range). Continuous data such as age, weight. duration of surgery, duration of anesthesia, awakening time, onset of agitation , duration of agitation, duration of PACU stay and PACU pain score were analyzed by unpaired Student's test. Categorical data such as gender , ASA physical status, a separation scale, an induction scale, type of operation, type of operation, an emergence agitation scale, intraoperative and PACU adverse events were compared using the Pearson's chi-square test. Incidence of emergence agitation and other adverse events were reported as number and percent (n, %). A P value of 0.05 was considered for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* children aged 1-9 years, with American Society of Anesthesiologists (ASA) physical status I or II ,
* scheduled to undergo elective ambulatory urologic surgery under general anesthesia combined with regional block

Exclusion Criteria:

* emergency procedures
* medical contraindication to placement of a caudal block
* mental retardation
* developmental delay
* attention-deficit/hyperactivity disorder
* psychiatric illness
* a history of paradoxical excitation with sedatives

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2010-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
the incidence of emergence agitation | average recovery room period was 120 minutes
  to compare the incidence of emergence agitation between sevoflurane anesthesia and desflurane anesthesia in pediatric ambulatory urologic surgery.

SECONDARY OUTCOMES:
the recovery profile | average recovery room period was 120 minutes
  to compare the recovery profile such as awakening time. Duration of PACU stay, and also intraopertive and PACU respiratory adverse events between sevoflurane anesthesia and desflurane anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Maliwan Oofuvong, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- Songklanagarind Hospital, Hat Yai, Changwat Songkhla, Thailand